CLINICAL TRIAL: NCT04255537
Title: Clinical Governance of Patients With Acute Coronary Syndrome in Italy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University Hospital of Ferrara (Other); AUSL Romagna Rimini (Other); Ospedale Morgagni-Pierantoni (Unknown); IRCCS Multimedica (Other); Azienda Usl di Bologna (Other Government); Ospedale Santa Maria delle Croci (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); ASST Cremona (Unknown)
Responsible Party: Principal Investigator, Sergio Leonardi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ESR-16-12480
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Myocardial Infarction; Quality Indicator; Percutaneous Coronary Intervention; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with STEACS intended for urgent angio/reperfusion.: This population mostly includes STEACS patients for whom primary PCI is intended. A minority of this population includes patients with STEACS intended for urgent angiography for persistent ST elevation and/or symptoms but with symptoms onset > 12 hours (secondary PCI), urgent angiography after failed fibrinolysis (rescue PCI), or patients receiving fibrinolysis.
- Patients with STEACS NOT intended for urgent angio/reperfusion: This population mostly includes STEACS patients not receiving reperfusion for late presentation (i.e. > 12 hours) or patient preference. Note that patient in this category may receive diagnostic angiography for better diagnostic assessment and/or risk stratification but NOT on an urgent basis.
- Patients with NSTEACS intended for invasive management: This population includes patients with NSTEACS managed invasively with coronary angiography within 72 hours. Most patients are a high-risk feature (i.e. positive troponin, GRACE risk score > 140, hemodynamic/electrical instability) for whom angiography is intended.
- Patients with NSTEACS NOT intended for invasive management: This population includes patients who are candidate for an initially conservative strategy. Note that this category may include patients who are subsequently managed with coronary angiography, including recurring symptoms of myocardial ischemia, or hemodynamic/ electrical instability.

SUMMARY:
This is a prospective, observational, multicenter study that enroll consecutive and all-comers patients hospitalized with a diagnosis of Acute Coronary Syndrome (ACS) at admission.

DETAILED DESCRIPTION:
This is a Quality Improvement Program which enroll all the consecutive patients hospitalized with ACS. The data elements that are central to the study include the primary and secondary quality indicators (QIs) that are used to define the performance and to promote improved quality of care.

At least 3000 patients will be enrolled. The primary endpoint are assessed in-hospital, at admission and discharge. Patients will be followed for 1 year after the ACS.

ELIGIBILITY:
Inclusion Criteria:

* STEACS patients: symptoms of myocardial ischemia and persistent (i.e. > 20 min) ST elevation in at least two contiguous ECG leads. N.B. Positive biomarkers of cardiac necrosis (i.e. troponin) are not required to confirm the diagnosis. New or presumably new left-bundle branch block at presentation occurs infrequently, may interfere with ST-elevation analysis, and should not be considered diagnostic of acute myocardial infarction (MI) in isolation.
* NSTE-ACS patients: symptoms of myocardial ischemia of at least 10 minutes without persistent ST elevation in at least two contiguous ECG leads. To be included in this category patients should have at least one of the following two conditions: a) ECG evidence of NSTEACS defined as T wave inversion in leads with dominant R waves of at least of at least 1 mm (100 μV) or ST segment depression of at least 0.5 mm (50 μV) and/or b) Biomarker evidence of NSTEACS defined as at least one positive (i.e. above the 99th percentile upper reference limit) troponin value (i.e. NSTEMI)
* A written informed consent (to agree for a contact, usually by telephone) is required only to patients who are discharged alive.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, are unable to comply with study follow up procedures, including, but not limited to, patients who are in prison, who are expected to move to a remote country, or who refuse to be followed should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed to include a consecutive and all-comers population hospitalized with a diagnosis of ACS at admission.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Time to reperfusion in patients with STEACS and optimal medical therapy at hospital discharge in patients with a final diagnosis of MI or UA. | Baseline

SECONDARY OUTCOMES:
To measure adherence to a wide range of QIs within multiple domains of care including optimal ACS diagnosis, therapy, and individualized risk assessment through monitoring of process of care measures and benchmarked quality-of-care feedback reports. | Baseline
Examine associations of program participation with trends of QIs adherence over 1 year. | 1 year.
To monitor the characteristics, treatments, and outcomes of patients hospitalized with ACS. | Baseline
To explore the association between evidence-based acute treatment strategies and risk-adjusted clinical outcomes. | 1 year.
To assess utilization of diagnostic imaging, laboratory tests and invasive procedures; and track hospital/coronary care unit length-of-stay data. | Baseline
Assess trends in medication dosing patterns, and improve drug safety through targeted quality feedback related to medication overdosing. | Baseline
Identify barriers to implementing guideline recommendations for patients with AMI, and develop effective strategies to overcome these barriers | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Leonardi, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (9):
- Italy (9):
  - Ferrara University Hospital, Cona, Ferrara
  - Ospedale Morgagni-Pierantoni, Forlì, Forlì-Cesena
  - IRCCS Multimedica, Sesto San Giovanni, Milano
  - Azienda Usl di Bologna, Bologna
  - ASST Cremona, Cremona
  - IRCCS Policlinico S. Matteo, Pavia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - AUSL Romagna, Rimini

REFERENCES:
- [Derived] Leonardi S, Montalto C, Carrara G, Casella G, Grosseto D, Galazzi M, Repetto A, Tua L, Portolan M, Ottani F, Galvani M, Gentile L, Cardelli LS, De Servi S, Antonelli A, De Ferrari GM, Visconti LO, Campo G; ACS Clinical Governance Programme Investigators. Clinical governance of patients with acute coronary syndromes. Eur Heart J Acute Cardiovasc Care. 2022 Nov 30;11(11):797-805. doi: 10.1093/ehjacc/zuac106. PMID 36124872
- [Derived] Leonardi S, Montalto C, Casella G, Grosseto D, Repetto A, Portolan M, Fortuni F, Ottani F, Galvani M, Cardelli LS, De Servi S, Rubboli A, De Ferrari GM, Oltrona Visconti L, Campo G. Clinical governance programme in patients with acute coronary syndrome: design and methodology of a quality improvement initiative. Open Heart. 2020 Dec;7(2):e001415. doi: 10.1136/openhrt-2020-001415. PMID 33372102